CLINICAL TRIAL: NCT05585619
Title: Difficult Encounters in a Chronic Pain Setting: An Analysis of Factors Associated With "Difficult"
Brief Title: Difficult Encounters in Pain Medicine
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00334965
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
Keywords: chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain patients: New chronic pain consults seen by a trainee and attending pain physician
  Interventions: Other: Pain treatment

INTERVENTIONS:
Other: Pain treatment — Any pain treatment to include medications, procedures, or referrals

SUMMARY:
The investigators are seeking to determine factors associated with difficult patient encounters in an academic pain clinic. The investigators are examining 36 different variables to determine the association with "difficult" patient encounters as independently rated by a trainee and attending physician.

DETAILED DESCRIPTION:
Pain is associated with significant psychosocial pathology include axis 1 diagnoses, opioid use and misuse, unemployment, and strained relationships, and treatments for chronic pain are often ineffective. Collectively, these factors may result in a higher prevalence of patients characterized as 'difficult', which can lead to missed diagnoses, barriers to care resulting in poorer outcomes (professional pessimism, mistrust, passive treatment, referrals to other providers or discharge), patient complaints and 'HERO' events, avoidable legal claims, and increased risk of professional burnout. Characterizing patients as "difficult" (instead of encounters) may have negative consequences for future care, and there are few studies that have explored patients' perspectives on "difficult" encounters. Although several articles have narratively explored this issue, there are few targeted at chronic pain patients, and no studies in this population that set out to determine what variables are associated with a "difficult encounter", the congruence between patients' and providers' impressions of an encounter, or whether difficult encounters are associated with pain treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Pain duration > 3 months
* New Visit (or no visit within 3 years)

Exclusion Criteria:

* Referral only for diagnostic procedure
* Friend or relative, or direct referral from friend or relative

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients seen for a new consultation at the Johns Hopkins Blaustein Pain Treatment Center
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Difficulty of encounter as rated by trainee | Immediately after consult
  Difficulty of encounter as rated by a 6-point Likert scale (1=very pleasant, 6=extremely difficult)
Difficulty of encounter as rated by attending physician | Immediately after consult
  Difficulty of encounter as rated by a 6-point Likert scale (1=very pleasant, 6=extremely difficult)

SECONDARY OUTCOMES:
Patient global impression of change | 1-2 months post-treatment
  1-7 Likert scale (1=no change or worse, 7=a great deal better)
Pain score | 1-2 months post-treatment
  0-10 numerical pain scale (0=no pain, 10= worst pain imaginable)
Categorical success | 1-2 months post-treatment
  Binary measure of success (2-point or greater decrease in average pain score coupled with a score of 5 or greater on Patient global impression of change scale)
Appointment status | 1-2 months post-treatment
  Showed up on time or showed up late or missed appointment
Number of side effects | 1-2 months post-treatment
  Side effects from medications or complications from procedures

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Variables studied, outcomes, statistical codes
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 1-3 years after completion of study
Access Criteria: By request

REFERENCES:
- [Result] Wasan AD, Wootton J, Jamison RN. Dealing with difficult patients in your pain practice. Reg Anesth Pain Med. 2005 Mar-Apr;30(2):184-92. doi: 10.1016/j.rapm.2004.11.005. PMID 15765460
- [Result] Hinchey SA, Jackson JL. A cohort study assessing difficult patient encounters in a walk-in primary care clinic, predictors and outcomes. J Gen Intern Med. 2011 Jun;26(6):588-94. doi: 10.1007/s11606-010-1620-6. Epub 2011 Jan 25. PMID 21264521
- [Derived] Liu WL, van Gelderen E, Mawalkar R, Wang EJ, Treisman G, Cohen SP. Do difficult encounters affect pain treatment outcomes? A prospective cohort study. Pain Med. 2025 Sep 1;26(9):554-561. doi: 10.1093/pm/pnaf027. PMID 40100641